CLINICAL TRIAL: NCT06953843
Title: An Umbrella Trial of Combining Different Radiotherapy Fractionation Patterns With Immunotherapy for Multiple Metastases of Non-Small Cell Lung Cancer
Brief Title: Study on the Optimal Combination Pattern of the Combined Treatment of Radiotherapy and Immunotherapy for the Abscopal Effect in Non-Small Cell Lung Cancer (NSCLC) With Multiple Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Prof, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-023
Record Dates: First submitted 2025-04-20; First posted 2025-05-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV Without EGFR/ALK Mutation
MeSH Terms: interventions — Drug Therapy; Radiotherapy; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental)
  Interventions: Drug: Benmelstobart combined with chemotherapy
- Group B (Experimental)
  Interventions: Drug: Benmelstobart combined with chemotherapy
- Group C (Experimental)
  Interventions: Drug: Benmelstobart combined with chemotherapy
- Group D (Experimental)
  Interventions: Drug: Benmelstobart combined with chemotherapy
- Group E (Experimental)
  Interventions: Drug: Benmelstobart combined with chemotherapy
- Group F (Experimental)
  Interventions: Drug: Benmelstobart combined with Bevacizumab and chemotherapy

INTERVENTIONS:
Drug: Benmelstobart combined with chemotherapy — After 4 cycles of treatment with Benmelstobart combined with chemotherapy, if there is no progression, the patient will receive the treatment of 6-10Gy*3-6F plus Benmelstobart.
  Other Names: Radiotherapy
  Arms: Group A
Drug: Benmelstobart combined with chemotherapy — After 4 cycles of treatment with Benmelstobart combined with chemotherapy, if there is no progression and the largest lesion measures between 3 cm and 5 cm, the patient will receive the treatment of 3 Gy * 15 fractions plus Benmelstobart.
  Other Names: Radiotherapy
  Arms: Group B
Drug: Benmelstobart combined with chemotherapy — After 4 cycles of treatment with Benmelstobart combined with chemotherapy, if there is no disease progression and the largest lesion is larger than 5 cm, the patient will receive treatment with Spatial Fractionated Radiotherapy Technique (SFRT) plus Benmelstobart.
  Other Names: Radiotherapy
  Arms: Group C
Drug: Benmelstobart combined with chemotherapy — After 4 cycles of treatment with Benmelstobart combined with chemotherapy, if there is no disease progression, and when the largest lesion is ≤ 3 cm and the patient can maintain the radiotherapy position for 50 minutes, the patient will receive treatment with the hyperfractionated pulsed radiotherapy technique (0.5 Gy * 16 * 6 fractions) plus Benmelstobart.
  Other Names: Radiotherapy
  Arms: Group D
Drug: Benmelstobart combined with chemotherapy — After 4 cycles of treatment with Benmelstobart combined with chemotherapy, Benmelstobart is continued for maintenance treatment.
  Arms: Group E
Drug: Benmelstobart combined with Bevacizumab and chemotherapy — For eligible subjects who have developed resistance to EGFR-TKI, after 4 cycles of treatment with Benmelstobart combined with Bevacizumab and chemotherapy, if there is no disease progression, they will receive the treatment of 6-10Gy * 3-6 fractions plus Benmelstobart.
  Other Names: Radiotherapy
  Arms: Group F

SUMMARY:
This study aims to conduct a prospective, multicenter, umbrella clinical study to compare the abscopal effects of different radiotherapy fractionation patterns combined with Benmelstobart, and to explore an efficient and low-toxic treatment strategy for non-small cell lung cancer (NSCLC) with multiple metastases. The main objective is to explore and compare the control rates of abscopal lesions in NSCLC patients with multiple metastases when different radiotherapy fractionation patterns are combined with Benmelstobart.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet all of the following inclusion criteria to be enrolled in this study:

  1. Non-small cell lung cancer confirmed by pathological histology.
  2. More than 3 metastatic lesions.
  3. No brain metastases or stable lesions.
  4. Negative for driver genes (including EGFR, ALK, ROS, BRAF, MET, RET).
  5. Performance status (PS) score of 0-1, with an expected survival period of more than 3 months.
  6. Age between 18 and 75 years old.
  7. Assessment by PET-CT (including FDG and FMISO, not mandatory).
  8. No contraindications to immunotherapy and radiotherapy.
  9. Signed the informed consent form.

Exclusion Criteria:

* Patients with any of the following criteria are not eligible for enrollment in this study:

  1. Those with severe dysfunction of important vital organs (heart, liver, kidney).
  2. Those accompanied by other malignant tumors.
  3. Uncontrolled heart diseases or myocardial infarction within the past 6 months.
  4. Those with a history of mental illness.
  5. Other situations in which the researcher deems it inappropriate for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2025-07-09 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The remission rate of abscopal lesions | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to approximately 2 years
  To evaluate the efficacy of Benmelstobart plus different radiotherapy fractionation modes in non-small cell lung cancer (NSCLC) patients with multiple metastases, as measured by the remission rate of abscopal lesions according to RECIST v1.1

SECONDARY OUTCOMES:
PFS | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to approximately 2 years
  To evaluate the efficacy of Benmelstobart plus different radiotherapy fractionation modes in non-small cell lung cancer (NSCLC) patients with multiple metastases, as measured by progression-free survival rate according to RECIST v1.1
OS | up to 5 years
  To evaluate the efficacy of Benmelstobart plus different radiotherapy fractionation modes in non-small cell lung cancer (NSCLC) patients with multiple metastases, as measured by by overall survival
AE | From date of consent informed until 60 days after the last investigational product administration. Up to approximately 2 years
  The incidence of immune-related adverse events (irAEs) as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Sun, MD, Principal Investigator — the second affiliated hospital of Army medical university, Chongqing, Chongqing 40037 Recruiting
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No